CLINICAL TRIAL: NCT02444624
Title: Clostridium and Neonatal Necrotizing Enterocolitis Pathophysiology : Clinical and Molecular Approaches
Acronym: CLOSNEC
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC14_0295
Record Dates: First submitted 2015-02-16; First posted 2015-05-14 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Necrotizing Enterocolitis
Keywords: necrotizing enterocolitis; Clostridium; premature birth
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- not necrotizing enterocolitis group: not necrotizing enterocolitis preterm neonates matched with necrotizing enterocolitis preterm neonates
- necrotizing enterocolitis group: necrotizing enterocolitis preterm neonates of gestational age less than or equal to 31+6 weeks of amenorrhoea with confirmed NEC diagnosis (Bell stage II or III)

SUMMARY:
The clinical study involves a French network of 20 neonatology centres created as part of the EPIFLORE project. Investigators propose including all premature babies with confirmed necrotizing enterocolitis (NEC) diagnosis (Bell stage II or III) paired with a control group of healthy premature babies, over a 2-year period. The clinical data will be entered at inclusion until departure from the department, and the ASQ (Ages and Stages Questionnaires) will be collected after 24 months. Samples from NEC cases and from the control group will be submitted for microbiological testing by culture and pyrosequencing. This will enable the main aerobic micro-organisms in the dominant and subdominant intestinal microbiota to be isolated. This case-control study will be used to compile a collection of clinical and microbiological data, in order to confirm the role of bacteria in the pathophysiology of NEC, and to confirm the involvement of bacteria from the Clostridium genus in particular.

DETAILED DESCRIPTION:
Necrotizing enterocolitis (NEC) remains an important cause of morbidity and mortality among preterm neonates. Despite many investigations its pathogenesis remains unclear. The role of intestinal bacteria in NEC development is supported by epidemiologic evidence (outbreaks), the frequent isolation of infectious agents, and a decrease incidence of NEC resulting from preventive antibiotic treatment. Bacterial implication is thought to be due to colonic fermentation of nonhydrolyzed lactose, a consequence of the intestinal immaturity of preterm infants (intestinal lactase deficiency). To date, no specific bacteria or bacterial colonization pattern have been causally associated with the development of NEC. Clinical signs and some epidemiological studies are consistent with clostridia involvement in NEC. Indeed, Clostridium butyricum, Clostridium perfringens, and Clostridium paraputrificum have been isolated from the blood, feces, and peritoneal fluids of preterm neonates suffering from NEC. In addition, a correlation between the presence of C. butyricum and C. paraputrificum and pneumatosis intestinalis in tissue specimens from NEC neonates was reported. Furthermore, the role of these clostridia species in NEC pathogenesis has been demonstrated using NEC animal models (preterm piglet or gnotobiotic quails). Particularly, lactose fermentation end-products (butyrate or iso-butyrate) was linked to cecal NEC-like lesions onset in gnotobiotic quails animal model.

This project is lying within this context, and aims at confirming the clostridial involvement in the pathogenesis of NEC and search for bacterial pathogenicity biomarkers. For this purpose, investigators will use both clinical and experimental approaches.

The clinical study will take the opportunity of previous EPIFLORE project network (ANR 2012) to build during a one-year period a large collection of proved NEC cases. During that period, preterm neonates diagnosed as NEC cases (Bell stage II or III) from 20 French neonatal units will be included and matched to a control group of non-NEC neonates. Anthropometric data, clinical data, drug and feeding intakes will be collected from birth to the neonatal unit discharge. Microbiota analysis of NEC and non-NEC preterm neonates will be performed using culture and 16S rRNA gene pyrosequencing. This case-control study aims at obtaining the largest French collection of clinical and microbiological documented NEC cases that will allow reaching significance in results about the characteristics of the microbiota of NEC neonates. Additionally, it will confirm the involvement of specific bacteria, i.e. clostridia, which will be proposed as a biological marker of high risk to develop NEC.

Experimental approach will consist in the construction of mutants of clinical isolates of C.butyricum, C. perfringens, and C. paraputrificum impaired in butyrate production using the Clostron directed mutagenesis knock out tool recently adapted to clostridia. investigators will inactivate the gene encoding the enzyme responsible for butyrate production. The pathogenicity of wild type and mutants strains will be performed in previous gnotobiotic quail animal model of NEC. This will allow us to verify the hypothesis of clostridia species biological involvement in NEC pathogenesis through fermentation end-product metabolite. This work will be completed by a phenotypic characterization and proteomics analysis of the clinical strains linked to NEC development in order to search for a bacterial pathogenicity biomarker. The absence of a consensus for the prevention of NEC is partly due to the lack of knowledge of its pathogenesis. This project will give important information in terms of clinical and mechanistic data. Looking for biological markers as investigators propose will be helpful for clinical practice and strategies of prevention implementation

ELIGIBILITY:
Inclusion Criteria "necrotizing enterocolitis group":

* Newborn gestational age less than or equal to 31 + 6 weeks of amenorrhea
* ECUN of diagnosis (Stage II or III Bell) confirmed
* Parental non-opposition / legal representative

Inclusion Criteria "not necrotizing enterocolitis group":

* Newborn gestational age less than or equal to 31 + 6 weeks of amenorrhea
* Respect for matching the order of priority set for criteria
* 1 of 2 control patients will be free of any antibiotic
* Parental non-opposition / legal representative

Exclusion criteria for both groups ("not necrotizing enterocolitis group" and "necrotizing enterocolitis group"): none

Max Age: 31 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Recruitment of CASES (NEC group) will prospectively occure according to the following schedule:
  Following the diagnosis confirmed ECUN (stage II or III Bell) during the stay in neonatology:
  * stool sample at the earliest
  * In case of surgery, if resection: a collection of intestinal contents and biopsy of the intestinal mucosa during the act
  * collection of clinical data from birth until hospital discharge or transfer of the child and then collecting the ASQ 24 months.
  Inclusion of control patients should be made within 7 days of the onset of the corresponding NEC case. Informed parents will previously allow enrollment of their child to set faeces sampling and data capture from birth to the output of hospitalization or transfer of the child and then collecting the ASQ 24 months.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2015-05-28 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2019-09-13 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the difference in prevalence of colonisation by bacteria from the Clostridium genus between the two study groups, CASE and CONTROL. | Inclusion until departure from hospital, an average of three months
  Results from analyses will not be used back for patients enrolled in this non interventional study

SECONDARY OUTCOMES:
Phenotypic comparison of clostridia between the 2 CASE and CONTROL groups | Inclusion until departure from hospital, an average of three months
  Results from analyses will not be used back for patients enrolled in this non interventional study

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Christophe Roze, Pr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes UH, Nantes, France